CLINICAL TRIAL: NCT06483113
Title: DAILIES TOTAL1® Soft Contact Lenses - Post-Market Clinical Follow-up Study
Status: Terminated | Type: Observational
Why Stopped: Management decision
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Other Study IDs: CLU484-N001
Record Dates: First submitted 2024-06-26; First posted 2024-07-03 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-07

CONDITIONS: Myopia; Hyperopia; Presbyopia; Astigmatism
Keywords: Contact lenses
MeSH Terms: conditions — Myopia; Hyperopia; Presbyopia; Astigmatism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (3):
- DAILIES TOTAL1 Sphere: Delefilcon A spherical soft contact lenses worn in both eyes in a real-world setting
  Interventions: Device: Delefilcon A spherical soft contact lenses
- DAILIES TOTAL1 Toric: Delefilcon A toric soft contact lenses worn in both eyes in a real-world setting
  Interventions: Device: Delefilcon A toric soft contact lenses
- DAILIES TOTAL1 Multifocal: Delefilcon A multifocal soft contact lenses worn in both eyes in a real-world setting
  Interventions: Device: Delefilcon A multifocal soft contact lenses

INTERVENTIONS:
Device: Delefilcon A spherical soft contact lenses — Silicone hydrogel contact lenses prescribed for single use, daily disposable wear (less than 24 hours while awake) for the correction of ametropia (myopia or hyperopia)
  Other Names: DAILIES TOTAL1® Spherical Contact Lenses
  Groups: DAILIES TOTAL1 Sphere
Device: Delefilcon A toric soft contact lenses — Silicone hydrogel contact lenses prescribed for single use, daily disposable wear (less than 24 hours while awake) for the correction of ametropia (myopia or hyperopia) with astigmatism
  Other Names: DAILIES TOTAL1® for Astigmatism Contact Lenses
  Groups: DAILIES TOTAL1 Toric
Device: Delefilcon A multifocal soft contact lenses — Silicone hydrogel contact lenses prescribed for single use, daily disposable wear (less than 24 hours while awake) for the correction of ametropia (myopia or hyperopia) with presbyopia
  Other Names: DAILIES TOTAL1® Multifocal Contact Lenses
  Groups: DAILIES TOTAL1 Multifocal

SUMMARY:
The purpose of this study is to continuously assess the visual performance and safety of DAILIES TOTAL1 soft contact lenses in a real world setting and broader patient base through routine clinical practices. This activity will be used to continuously support delefilcon A (sphere, toric, and multifocal) soft contact lens regulatory requirements and standards.

DETAILED DESCRIPTION:
This study includes a Baseline visit and a Year 1 visit.

The Baseline visit is defined as the first office visit where an eye care professional provided an in-person office biomicroscopy exam to the subject before or during which a DAILIES TOTAL1 sphere, toric, or multifocal soft contact lens prescription was released. The Baseline visit will be retrospective. All assessments at baseline will be obtained from chart reviews.

The Year 1 visit is defined as the visit that occurs 1 year (-2/+4 months) since the Baseline visit during which period the subject is wearing prescribed lenses and a contact lens examination is performed. The Year 1 visit can be either retrospective or prospective in subjects 7 to less than 18 years of age. For subjects 18 years of age and older, the Year 1 visit will be retrospective.

ELIGIBILITY:
Key Inclusion Criteria:

* At baseline: 7 years of age or older for sphere and toric wearers, 40 years of age or older for multifocal wearers.
* Wearers of delefilcon A (sphere, toric, or multifocal) soft contact lenses of the same design in both eyes who have already begun use of the lens type and have purchased at least 3-month supply of lenses at baseline.
* Best corrected distance visual acuity (BCVA) 20/25 or better in each eye at baseline.
* Other protocol-defined inclusion criteria may apply.

Key Exclusion Criteria:

* Any ocular disease or condition that would contraindicate contact lens wear at baseline.
* Use of systemic or ocular medications that would contraindicate contact lens wear at baseline.
* Other protocol-defined exclusion criteria may apply.

Min Age: 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Subjects will be recruited from clinical sites located in the United States.
Sampling Method: Non-Probability Sample
Enrollment: 192 (Actual)
Dates: Start 2024-11-26 (Actual); Primary Completion 2025-02-27 (Actual); Study Completion 2025-02-27 (Actual)

PRIMARY OUTCOMES:
Distance visual acuity (VA) with study lenses at Baseline - Sphere and Toric | Baseline
  Distance VA will be assessed for each eye individually with study lenses in place and recorded in Snellen. This endpoint is prespecified for DAILIES TOTAL1 spherical contact lenses and DAILIES TOTAL1 for Astigmatism contact lenses.
Distance visual acuity with study lenses at Year 1 Follow-up - Sphere and Toric | Year 1 Follow-Up
  Distance VA will be assessed for each eye individually with study lenses in place and recorded in Snellen. This endpoint is prespecified for DAILIES TOTAL1 spherical contact lenses and DAILIES TOTAL1 for Astigmatism contact lenses.
Distance visual acuity with study lenses at Baseline - Multifocal | Baseline
  Distance visual acuity will be assessed for both eyes together with study lenses in place and recorded in Snellen. This endpoint is prespecified for DAILIES TOTAL1 multifocal contact lenses.
Distance visual acuity with study lenses at Year 1 Follow-Up - Multifocal | Year 1 Follow-Up
  Distance visual acuity will be assessed for both eyes together with study lenses in place and recorded in Snellen. This endpoint is prespecified for DAILIES TOTAL1 multifocal contact lenses.
Near visual acuity with study lenses at Baseline - Multifocal | Baseline
  Near visual acuity will be assessed for both eyes together with study lenses in place and recorded in Snellen. This endpoint is prespecified for DAILIES TOTAL1 multifocal contact lenses.
Near visual acuity with study lenses at Year 1 Follow-Up - Multifocal | Year 1 Follow-Up
  Near visual acuity will be assessed for both eyes together with study lenses in place and recorded in Snellen. This endpoint is prespecified for DAILIES TOTAL1 multifocal contact lenses.
Incidence of corneal infiltrative events | Up to Year 1
  A corneal infiltrate is a single or group of inflammatory cells in the normally clear cornea.
Incidence of microbial keratitis | Up to Year 1
  Microbial keratitis is a sight-threatening infection of the cornea.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Lead, Vision Care, Study Director — Alcon Research, LLC
Locations (12):
- United States (12):
  - Westview Optometry, San Diego, California
  - Scripps Optometric Group, San Diego, California
  - Dr. Walker and Associates, Ponte Vedra Beach, Florida
  - Advanced Eyecare Specialists, West Palm Beach, Florida
  - The Eye Doctors Inc, Eden Prairie, Minnesota
  - Cornea and Contact Lens Institute of Minnesota, Edina, Minnesota
  - Complete Eye Care of Medina, Medina, Minnesota
  - Koetting Associates, St Louis, Missouri
  - Center for Ophthalmic and Vision Research, New York, New York
  - Optometry Group, PLLC, Memphis, Tennessee
  - Southern Utah Medical Research, St. George, Utah
  - Spokane Eye Clinic, Spokane, Washington

IPD SHARING:
Plan to Share IPD: No